CLINICAL TRIAL: NCT05891028
Title: 64Cu/68Ga Labelled EB-ss-CPT PET/CT Scan in Colorectal Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-EB-CPT
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; PET/CT; CPT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-EB-ss-CPT PET/CT scan (Experimental): 68Ga-EB-ss-CPT PET/CT scan Dosimetry study about 6 patients were injected with 3 (MBq) per kilogram body weight of 68Ga-EB-ss-CPT PET/CT in one dose intravenously and underwent wholebody scan at 5min#30min#60min#120min#240min, then analysis of dosimetric distribution ofradiopharmaceuticals in human body by HERMES software.
  Interventions: Drug: 68Ga-EB-ss-CPT
- 64Cu-EB-ss-CPT PET/CT scan (Experimental): 64Cu-EB-ss-CPT PET/CT scan Dosimetry study about 6 patients were injected with 2 (MBq) per kilogram body weight of 64Cu-EB-ss-CPT PET/CT in one dose intravenously and underwent wholebody scan at 30min#8h#12h#24h#48h, then analysis of dosimetric distribution ofradiopharmaceuticals in human body by HERMES software.
  Interventions: Drug: 64Cu-EB-ss-CPT

INTERVENTIONS:
Drug: 68Ga-EB-ss-CPT — 68Ga-EB-ss-CPT were intravenous injected into the patients before PET/CT scans
  Other Names: 68Ga
  Arms: 68Ga-EB-ss-CPT PET/CT scan
Drug: 64Cu-EB-ss-CPT — 64Cu-EB-ss-CPT were intravenous injected into the patients before PET/CT scans
  Other Names: 64Cu
  Arms: 64Cu-EB-ss-CPT PET/CT scan

SUMMARY:
Positron labeled camptothecin based PET imaging is a new imaging technique that uses positron isotopes such as 68Ga/64Cu for PET/CT (MR) imaging. It is expected to have significant clinical significance in staging and detecting primary and metastatic head and neck cancer, oral cancer, and colorectal cancer tumors.

DETAILED DESCRIPTION:
CPT, a botanical anticancer drug, is a mechanism that inhibits DNA synthesis and thus exerts anticancer effects by using topoisomerase I as its target of action, and has shown good efficacy in digestive system tumors and head and neck tumors, etc. Previous research result showed that amphiphilic EB-ss-CPT formed nanoparticles by self-assembly, bound to albumin in vivo and released CPT by breaking disulfide bonds under high GSH conditions in tumor tissues, effectively enhancing the pharmacokinetics and biodistribution of camptothecin, thereby improving therapeutic efficacy and In this study, the sensitivity of colorectal cancer cells to the drug was also demonstrated. In this study, 64Cu-NOTA-EB-ss-CPT (hereafter 64Cu-EB-CPT) was generated by posionuclide 64Cu-labelled EB-ss-CPT for PET/CT imaging alone and showed better tumour enrichment compared to the 64Cu-labelled CPT group. EB-CPT is expected to be more enriched in tumour tissue through the EPR effect of its nanoparticles, and 64Cu is also a promising radionuclide for quantitative analysis using PET/CT imaging. The formation of 64Cu-EB-CPT or 68Ga-EB-CPT by labelling EB-CPT with the positronium nuclide 64Cu or 68Ga is expected to be enhanced by the EPR effect of the precursors (the enhanced permeability and retention effect of solid tumours). The EPR effect (enhanced permeability and retention effect) refers to the tendency of molecules or particles of certain sizes to accumulate in tumour tissue relative to normal tissue) is expected to enrich the drug in the tumour area and allow early diagnosis of tumour patients by PET/CT imaging with the preceding positronuclide 64Cu or 68Ga, which can help in the staging of tumours and the development of treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* In the near future (within 2 months), patients who plan to undergo puncture biopsy or undergo tumor surgical treatment or are clinically highly suspected of cancer (including primary and tumor recurrence and metastasis)
* Able to understand and voluntarily sign informed consent forms, with good compliance

Exclusion Criteria:

* Severe abnormalities in liver and kidney function
* Suffering from claustrophobia or other mental illnesses
* Pregnant, pregnant, and lactating women

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Dosimetric distribution of radiopharmaceuticals | 2 months
  Input the data of 5-6 patients into HERMES software, and analyze the dose distribution of radioactive drugs in human body through HERMES software
Standardized uptake value | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast tumor will be measured. SUV were obtained by a self-made software and referring to phantom study.If the SUV value cannot be obtained, the COUNTS of target organ/background ratio between the lesion and surrounding tissues shall be used for calculation.

SECONDARY OUTCOMES:
Adverse events collection | 1 year
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Science & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China